CLINICAL TRIAL: NCT04520126
Title: Effect of Olivomed (Olive Extract) on Endothelial, Cardiac and Vascular Function of Patients With Stable Coronary Artery Disease
Brief Title: Effect of Olivomed (Olive Extract) on Endothelial, Cardiac and Vascular Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor of Cardiology, University of Athens
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Oliveheart
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
Keywords: olive oil, myocardial deformation, glycocalyx
MeSH Terms: conditions — Coronary Artery Disease | interventions — 3,4-dihydroxyphenylethanol; oleocanthal

STUDY DESIGN:
Intervention Model Description: 30 patients will be randomized to Olivomed (5 mg hydroxytyrosol po twice daily) or placebo for one month and then they will be crossed over to the alternate treatment for another one month.
  30 patients will be randomized to OlivomedSmart ((OL:HT:OC 2:1:3) - 5 mg hydroxytyrosol po twice daily) or placebo for one month and then they will be crossed over to the alternate treatment for another one month.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- olive extract 1 - olivomed (Active Comparator): 15 patients will be randomized to receive two Olivomed soft capsules bid for one month (5 mg hydroxytyrosol po twice daily) and then they will be crossed over to treatment placebo for another one month.
  Interventions: Dietary Supplement: Olivomed (capsules containing hydroxytyrosol); Dietary Supplement: OlivomedSmart - Capsules containing - combination of Oleuropein (OL), Hydroxytyrosol (HT), Oleocanthal (OC) - (OL:HT:OC 2:1:3), (5 mg HT bid).
- placebo 1 (Placebo Comparator): 15 patients will be randomized to receive two placebo soft capsules bid for one month. Then they will be crossed over to receive two Olivomed soft capsules bid for oen month (5 mg hydroxytyrosol po twice daily)
  Interventions: Dietary Supplement: Olivomed (capsules containing hydroxytyrosol); Dietary Supplement: OlivomedSmart - Capsules containing - combination of Oleuropein (OL), Hydroxytyrosol (HT), Oleocanthal (OC) - (OL:HT:OC 2:1:3), (5 mg HT bid).
- olive extract 2 - olivomedSmart (Active Comparator): 15 patients will be randomized to receive two soft capsules containing OL:HT:OC (2:1:3) bid for one month (5 mg hydroxytyrosol po twice daily) and then they will be crossed over to treatment placebo for another one month.
  Interventions: Dietary Supplement: Olivomed (capsules containing hydroxytyrosol); Dietary Supplement: OlivomedSmart - Capsules containing - combination of Oleuropein (OL), Hydroxytyrosol (HT), Oleocanthal (OC) - (OL:HT:OC 2:1:3), (5 mg HT bid).
- placebo2 (Placebo Comparator): 15 patients will be randomized to receive two placebo soft capsules bid for one month. Then they will be crossed over to receive two soft capsules containing OL:HT:OC (2:1:3) bid for one month (5 mg hydroxytyrosol po twice daily) bid for one month.
  Interventions: Dietary Supplement: Olivomed (capsules containing hydroxytyrosol); Dietary Supplement: OlivomedSmart - Capsules containing - combination of Oleuropein (OL), Hydroxytyrosol (HT), Oleocanthal (OC) - (OL:HT:OC 2:1:3), (5 mg HT bid).

INTERVENTIONS:
Dietary Supplement: Olivomed (capsules containing hydroxytyrosol) — patients with stable coronary artery disease will be randomised to Olivomed or placebo for one month and then they will be crossed over to the alternate treatment for one month.
  Other Names: placebo soft capsules
Dietary Supplement: OlivomedSmart - Capsules containing - combination of Oleuropein (OL), Hydroxytyrosol (HT), Oleocanthal (OC) - (OL:HT:OC 2:1:3), (5 mg HT bid). — patients with stable coronary artery disease will be randomised to combination of OL, HT, OC or placebo for one month and then they will be crossed over to the alternate treatment for one month.
  Other Names: placebo soft capsules

SUMMARY:
Olive extracts are considered to have antioxidant properties. The investigators will study the effect of olive extracts containing hydroxytyrosol (HT)-olivomed and combination of Oleuropein (OL), Hydroxytyrosol (HT), Oleocanthal (OC) - olivomedSmart on endothelial, cardiac and vascular function in patients with coronary artery disease .

DETAILED DESCRIPTION:
30 patients with stable angiographically documented coronary artery disease will be randomized to receive olive extracts with high concentration of hydroxytyrosol (5 mg po twice per day included in Olivomed capsules) or placebo for one month and then they will be switched off to the alternate treatment (placebo or Olivomed capsules) for another one month.

30 patients with stable angiographically documented coronary artery disease will be randomized to receive OlivomedSmart - olive extracts with Oleuropein (OL), Hydroxytyrosol (HT), Oleocanthal (OC) (OL:HT:OC 2:1:3) or placebo for one month and then they will be switched off to the alternate treatment (placebo or Olivomed capsules) for another one month.

the same quantity of hydroxytyrosol was contained in two supplements.

ELIGIBILITY:
Inclusion Criteria:

1. Age <70 years
2. Stable coronary heart disease
3. Patients with acute coronary syndrome who have undergone percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), 2 months must have passed since the incident
4. High LDL levels, low HDL, high triglycerides

Exclusion Criteria:

1. Age> 70 years
2. Patient with diabetes
3. Patient with hypertension
4. Patient with liver disease
5. Patient with thyroid disease
6. Patient with active malignancy
7. Patient with a disease that affects inflammatory markers (rheumatic diseases, etc.)
8. Patient with chronic renal failure (creatinine> 2 mg / dl)
9. Patient treated chronically with corticosteroids
10. Patient who has joined a weight loss program or any dietary intervention or intensive exercise programme within the previous 2 months or consumes multivitamin preparations with antioxidant properties.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Olivomed and OlivomedSmart effects on endothelial glycocalyx thickness. | one month
  Olivomed and OlivomedSmart effects on endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels using Sidestream Darkfield (SDF) imaging
Olivomed and OlivomedSmart effects on endothelial function. | one month
  Olivomed and OlivomedSmarteffects on endothelial function. Endothelial function is assessed by measuring Flow Mediated Vasodilation (FMD) of the brachial artery using ultrasonography. During FMD test, vasodilation occurs following an acute increase in blood flow, typically induced via circulatory arrest in the arm (supra-systolic cuff occlusion) for 5 minutes. FMD is the percent of increase of the brachial artery diameter during hyperemia after release of the occlusion.
Olivomed and OlivomedSmart effects on arterial stiffness | one month
  Olivomed and OlivomedSmart effects on on arterial stiffness as assessed by carotid to femoral pulse wave velocity (PWV, m/s) using tonometry.
Olivomed and OlivomedSmarteffects on coronary function. | one month
  Olivomed and OlivomedSmart effects on coronary function as assessed by measuring coronary flow reserve of Left anterior descending artery. Coronary flow reserve is estimated by Doppler echocardiography as the ratio of coronary flow velocity after bolus intravenous adenosine infusion to coronary flow velocity at rest.
Olivomed and OlivomedSmart effects on left ventricular function. | one month
  Olivomed and OlivomedSmart effects on left ventricular function as assessed by Global Longitudinal Strain using speckle tracking echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Principal Investigator — 2nd Cardiology Department, National and Kapodistrian University of Athens, Attikon General Hospital
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece